CLINICAL TRIAL: NCT03679520
Title: Antenatal Preparation for Early Parenthood: A Pilot Study of a Cluster Randomised Controlled Trial Evaluating a New Programme Based on First-time Parents' Preferences
Brief Title: New Programme for Antenatal Preparation for Early Parenthood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2017/746
Record Dates: First submitted 2018-09-03; First posted 2018-09-20 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Parents
Keywords: Prenatal education; Parents; Randomized controlled trial; Self Efficacy; Depression, postpartum
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: Antenatal clinics randomised to control group provide antenatal parental preparation as usual (regular programme) to expectant parents and antenatal clinics randomised to intervention group provide a new programme of antenatal parental preparation to expectant parents.
Who Masked: Participant
Masking Description: Individual participant information will state that different ways of providing antenatal parental preparation will be evaluated, but will not reveal any specific information about the different types of antenatal parental preparation. Individual participants will therefore have no knowledge of allocation to control group or intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New programme (Experimental): A new programme of antenatal parental preparation provided by midwives to groups with 8-16 individuals. It will include 5 sessions á 2 hours and start in gestational week 25.
  Interventions: Other: New programme
- Regular programme (Active Comparator): A regular programme of antenatal parental preparation provided by midwives to groups of 8-16 individuals and encompassing between 5 and 7 hours of antenatal parental preparation.
  Interventions: Other: Regular programme

INTERVENTIONS:
Other: New programme — Time for topics related to the time after birth and in reversed chronological order to give an early and joint focus on parenthood for both parents. Involving new parents to share their experiences of early parenthood with expectant parents. Introducing and using evidence-based websites in the sessions A breastfeeding preparation that gives tools to meet common challenges in the initial phase of breastfeeding. Based on principles for adult learning.
  Sessions
  1. Introduction, life-change of becoming a parent and co-parenting
  2. Early parenthood
  3. Breastfeeding, caring for the baby and early parenthood
  4. and 5 Labour, birth and postnatal care
  Arms: New programme
Other: Regular programme — Antenatal parental preparation "as usual". As no guidelines exist the number of sessions may vary between 2 and 3 sessions and smaller variations in content may also occur.
  Sessions
  1. (or 1 and 2) Labour, birth and postnatal care
  2. or 3 Breastfeeding, caring for the baby and early parenthood
  Arms: Regular programme

SUMMARY:
Becoming a parent is a challenging stage in life, which provokes feelings of both excitement and insecurity; parents strive to develop confidence in their parenting role. Studies show that new parents often feel inadequately prepared for early parenthood which may have a negative impact on adjustment to life as a parent as well as health and wellbeing for the whole family.

The overall aim is to develop, pilot test and evaluate a new programme for antenatal preparation for the early parenthood period. The hypothesis is that expectant first-time parents who receive an intervention with a new programme for antenatal preparation for parenthood will show higher scores for parental self-efficacy in the early parenthood period than those who do not receive the intervention. The specific aims for the pilot study are:

1. To assess the acceptability of the procedures for parents and providers (midwives)
2. To estimate the likely rates of recruitment and retention of participants
3. To estimate the effects on outcome measurements in order to calculate the appropriate sample size in a full scale randomized controlled trial (RCT).

Antenatal clinics will be randomised to either intervention group, and provide a new programme of antenatal parental preparation, or to control group and provide a regular programme of antenatal parental preparation. First-time expectant parents will be invited in early pregnancy by the midwives at the antenatal clinics to participate in the study by partaking in an evaluation of the different ways to provide antenatal parental preparation. Parents who agree to participate will receive postal questionnaires before the antenatal parental preparation start and approximately four weeks after giving birth.

Midwives working in antenatal clinics randomised to the intervention group will receive a one-day-education before providing the intervention antenatal parental preparation. These midwives will also receive questionnaires, after the education and after providing the antenatal parental preparation.

All midwives, in both control group and intervention group, providing antenatal parental preparation will be given a form with questions related to the content in the provided programme to fill in.

DETAILED DESCRIPTION:
Development of the intervention; The development of the intervention was guided by the Medical Research Council's (MRC) framework for development and evaluation of complex interventions. The development phase involves identifying the evidence base, identifying or developing theory and modelling process and outcome. Based on reviews of literature and the results of previous studies in this project, the concept of self-efficacy in Social Cognitive Theory was identified as a suitable theory in the development and evaluation of the intervention.

Details of recruitment and randomisation of Antenatal clinics; Antenatal clinics (ANCs), which offer the most common model (regular) for antenatal parental preparation, as mapped out in a previous study, will be invited to participate in the pilot study which will compare the regular programme for antenatal parental preparation (control group) with a new programme for antenatal parental preparation (intervention group). Cluster randomisation of ANCs will be used to minimise contamination between the different programmes of antenatal preparation in the two groups. Randomisation will be stratified according to Care Need Index (CNI) which is based on socio-demographic variables of expectant mothers registered with the participating ANCs. A mean value of the CNIs of participating ANCs will be calculated, those below the mean value will form one strata and those above the mean value will form the other strata. Half of the ANCs will be randomised to the intervention group and half to the control group.

Details of preparations to provide the new programme intervention; A full-day education will be provided for midwives at the ANCs randomised to the intervention group which will include group leadership skills to facilitate peer learning among parents, evidence-based websites, framework for co-parenting and details regarding the new programme. The education to the midwives will be followed up with personal phone contact 1-2 months after the education, by the educator, in order to give opportunities for questions and clarifications in order to provide the intervention programme.

ELIGIBILITY:
Inclusion Criteria:

* Expectant first-time parents
* Intention to participate in group based antenatal parental preparation
* Understand written and spoken Swedish

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
The Parent Expectations Survey | 4 weeks postnatal
  The Parent Expectation Survey (PES) will be used to assess parental self-efficacy. PES exists in two versions, one for prenatal use and one for postnatal use. Both versions contain 25 items with statements related to their perceived parental skills, the phrasing of the statements in the prenatal version is prefaced with "I will…" and in the postnatal version "I can…" otherwise the statements are identical. The statements are answered on 11-point Likert-type scales ranging from 0 (Cannot do) to 10 (Certain can do). Total score range 0-250. Higher scores indicate higher parental self-efficacy. Statistical comparison will be made to assess the change of parental self-efficacy (total score) across time, from baseline to postnatal follow-up, and groups.

SECONDARY OUTCOMES:
The Parents' Postnatal Sense of Security Instrument | 4 weeks postnatal
  The Parents Postnatal Sense of Security (PPSS) will be used to assess parental sense of security during the early postnatal period. PPSS exists in two versions, one for mothers and one for partners. Mothers' version contain 18 items within 4 dimensions, partners' version 13 items within 4 dimensions, answered on 4-point Likert-type scales (1-4)
  Mothers' version: total score range 18-72. Dimensions: a sense of the midwives'/nurses' empowering behaviour 6-24; a sense of general well-being 5-20; a sense of afﬁnity within the family 4-16; and a sense that breast feeding was manageable 3-12.
  Partners': total score range 13-52. Dimensions: a sense of the midwives/nurses' empowering behaviour 5-20; a sense of the mother's general well-being including breastfeeding 3-12; a sense of general well-being 3-12; and a sense of afﬁnity within in the family 2-8.
  Higher scores indicate higher sense of security. Statistical comparisons will be made at dimension levels and the total score level
The Edinburgh Postnatal Depression Scale | 4 weeks postnatal
  The Edinburgh Postnatal Depression Scale (EPDS) will be used to assess risk of postnatal depression. EPDS is a 10-item self-report scale specifically designed to screen for postnatal depression in community samples. Each item is scored on a four-point scale (score 0-3), the total score range is 0-30. The risk for postnatal depression increases as scores increase. Statistical comparisons will be made at the total score level.

CONTACTS AND LOCATIONS:
Overall Officials: Linda J Kvist, PhD, Study Chair — Lund University
Locations (7):
- Sweden (7):
  - Barnmorskemottagningen Dalby, Dalby
  - Barnmorskorna Mitt i Skåne, Höör
  - Barnmorskemottagningen Kävlinge, Kävlinge
  - Barnmorskemottagningen Knislinge, Knislinge
  - Barnmorskemottagningen Capio Singelgatan, Malmo
  - Barnmorskemottagningen Capio Västra hamnen, Malmo
  - Barnmorskemottagningen Granen, Malmo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reece SM. The parent expectations survey: a measure of perceived self-efficacy. Clin Nurs Res. 1992 Nov;1(4):336-46. doi: 10.1177/105477389200100404. PMID 1483137
- [Background] Persson EK, Fridlund B, Dykes AK. Parents' postnatal sense of security (PPSS): development of the PPSS instrument. Scand J Caring Sci. 2007 Mar;21(1):118-25. doi: 10.1111/j.1471-6712.2007.00442.x. PMID 17428223
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Background] MRC (2006). Developing and evaluating complex interventions: new guidance. Medical Research Council. Available [2018-08-28] at https://www.mrc.ac.uk/documents/pdf/complex-interventions-guidance/
- [Background] Entsieh AA, Hallstrom IK. First-time parents' prenatal needs for early parenthood preparation-A systematic review and meta-synthesis of qualitative literature. Midwifery. 2016 Aug;39:1-11. doi: 10.1016/j.midw.2016.04.006. Epub 2016 Apr 28. PMID 27321714
- [Background] Palsson P, Persson EK, Ekelin M, Kristensson Hallstrom I, Kvist LJ. First-time fathers experiences of their prenatal preparation in relation to challenges met in the early parenthood period: Implications for early parenthood preparation. Midwifery. 2017 Jul;50:86-92. doi: 10.1016/j.midw.2017.03.021. Epub 2017 Mar 31. PMID 28399472
- [Background] Palsson P, Kvist LJ, Ekelin M, Hallstrom IK, Persson EK. "I Didn't Know What to Ask About": First-Time Mothers' Conceptions of Prenatal Preparation for the Early Parenthood Period. J Perinat Educ. 2018 Jun;27(3):163-174. doi: 10.1891/1058-1243.27.3.163. PMID 30364409
- [Background] Feinberg ME. Coparenting and the transition to parenthood: a framework for prevention. Clin Child Fam Psychol Rev. 2002 Sep;5(3):173-95. doi: 10.1023/a:1019695015110. PMID 12240706
- [Background] Bandura, A. (1997). Self-efficacy: the exercise of control. New York: W. H. Freeman and Company.
- [Background] Barimani M, Vikstrom A, Rosander M, Forslund Frykedal K, Berlin A. Facilitating and inhibiting factors in transition to parenthood - ways in which health professionals can support parents. Scand J Caring Sci. 2017 Sep;31(3):537-546. doi: 10.1111/scs.12367. Epub 2017 Jan 31. PMID 28144992
- [Background] Svensson J, Barclay L, Cooke M. Randomised-controlled trial of two antenatal education programmes. Midwifery. 2009 Apr;25(2):114-25. doi: 10.1016/j.midw.2006.12.012. Epub 2007 Apr 24. PMID 17459542